CLINICAL TRIAL: NCT04212832
Title: Transmuscular Quadratus Lumborum Block Block for Congenital Hip Dislocation Surgery: Randomized Controlled Study
Brief Title: Quadratus Lumborum Block for Congenital Hip Dislocation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTFANESTHESIAHIPQLB
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Congenital Hip Dislocation
MeSH Terms: conditions — Hip Dislocation, Congenital | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided quadratus lumborum block (Active Comparator): ultrasound guided quadratus lumborum block with 0.5 ml/kg % 0.25 bupivacaine
  Interventions: Drug: Bupivacaine
- No intervention (Other): Standard Pain Followup and Monitorization
  Interventions: Other: Standard pain

INTERVENTIONS:
Drug: Bupivacaine — 0.5 ml/kg %0.25 bupivacaine
  Arms: ultrasound guided quadratus lumborum block
Other: Standard pain — Standard pain follow up and monitorization
  Arms: No intervention

SUMMARY:
Developmental dysplasia of the hip (DDH) is one of the major disorder of the pediatric population with an incidence of 3 to 5 per 1000 children. Open surgical reduction of congenital hip dislocation (CHD) is typically performed after an ineffective closed reduction or older than 18 months. Multiple femoral or pelvic osteotomies and tenotomies are performed during this surgical treatment and cause severe postoperative pain.Since initial description for abdominal surgery, the quadratus lumborum block has experienced several surgeries for postoperative pain management in adults and pediatrics. One of these indication is the hip surgery and described for adult hip arthroplasty. In addition we reported two pediatric cases that single dose transmuscular quadratus lumborum block is an affective analgesia for CHD surgery. The aim of this study was to evaluate the analgesic effect of ultrasound guided transmuscular quadratus lumborum block in pediatric patients undergoing CHD surgery.

ELIGIBILITY:
Inclusion Criteria:

- American Society of Anesthesiologist's physiologic state I-II patients undergoing hip dislocation surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases
* Incomplete patient forms
* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* American Society of Anesthesiologist's III-IV

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability Score (FLACC) | Postoperative first 24hour
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Need for rescue analgesic | 2 hour
  Number of patients who required rescue analgesia in postoperative care unit in the first 2 hour
Need for analgesic | 24 hour
  Number of patients who required analgesic in the first 24 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahiskalioglu A, Yayik AM, Alici HA, Ezirmik N. Ultrasound guided transmuscular quadratus lumborum block for congenital hip dislocation surgery: Report of two pediatric cases. J Clin Anesth. 2018 Sep;49:15-16. doi: 10.1016/j.jclinane.2018.05.018. Epub 2018 May 26. No abstract available. PMID 29807213
- [Background] Ahiskalioglu A, Yayik AM, Alici HA. Response to Ince et al.: Ultrasound-guided quadratus lumborum plane block for congenital hip dislocation surgery: Dermatomes and osteotomes 'J Clin Anesth. 2018;54:140'. J Clin Anesth. 2019 Sep;56:39-40. doi: 10.1016/j.jclinane.2019.01.022. Epub 2019 Jan 23. No abstract available. PMID 30684924
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Celik EC. [Continuous quadratus lumborum type 3 block provides effective postoperative analgesia for hip surgery: case report]. Braz J Anesthesiol. 2019 Mar-Apr;69(2):208-210. doi: 10.1016/j.bjan.2018.06.007. Epub 2018 Sep 6. PMID 30195631
- [Background] Tulgar S, Ermis MN, Ozer Z. Combination of lumbar erector spinae plane block and transmuscular quadratus lumborum block for surgical anaesthesia in hemiarthroplasty for femoral neck fracture. Indian J Anaesth. 2018 Oct;62(10):802-805. doi: 10.4103/ija.IJA_230_18. PMID 30443064